CLINICAL TRIAL: NCT00589056
Title: A Phase I/II Trial of Protease Inhibitor, Nelfinavir, Given With Concurrent Thoracic Chemoradiotherapy in Patients With Locally-Advanced Non-Small Cell Lung Cancer
Brief Title: Nelfinavir, Radiation Therapy, Cisplatin, and Etoposide in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04507; IRB-806285; CDR0000582319
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Nelfinavir; Immunohistochemistry; Biopsy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Nelfinavir
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: nelfinavir mesylate; Genetic: protein expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Drug: nelfinavir mesylate
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Nelfinavir may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells. Nelfinavir may make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving nelfinavir together with radiation therapy, cisplatin, and etoposide may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of nelfinavir when given together with radiation therapy, cisplatin, and etoposide and to see how well they work in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose-limiting toxicities, maximum tolerated dose, and recommended phase II dose of nelfinavir mesylate when administered in combination with concurrent thoracic radiotherapy, cisplatin, and etoposide in patients with unresectable locally advanced non-small cell lung cancer.

Secondary

* To determine the tumor response at 3 months after completion of treatment as measured by RECIST criteria.
* To assess the inhibition of p-Akt in primary tumor or pathologic lymph nodes and in peripheral blood lymphocytes after 5-10 days of treatment with nelfinavir mesylate.
* To determine the median overall survival (OS) of patients treated with this regimen.
* To compare the observed median OS of these patients with the historical median OS of 17 months.

OUTLINE: This is a phase I, dose-escalation study of nelfinavir mesylate followed by a phase II study.

* Phase I: Patients receive oral nelfinavir mesylate twice daily beginning 1-2 weeks before the initiation of chemoradiotherapy and continuing until the completion of radiotherapy. Patients undergo thoracic radiotherapy once daily 5 days a week for 7-8 weeks. Patients also receive cisplatin IV on days 1, 8, 29, and 36 and etoposide IV on days 1-5 and 29-33. After completion of chemoradiotherapy, patients receive two additional courses of cisplatin and etoposide.
* Phase II: Patients receive nelfinavir mesylate at the maximum tolerated dose determined in phase I and concurrent chemoradiotherapy as in phase I.

Patients undergo blood sample collection periodically for correlative laboratory studies. Patients treated in the phase II portion of the study and those with primary tumors or pathologic lymph nodes easily accessible by core biopsy or mediastinoscopy also undergo tumor tissue biopsies. Blood and tumor tissue samples are analyzed for expression of molecular markers (total Akt and p-Akt ) by immunohistochemistry. The molecular markers are correlated with treatment response.

After completion of study treatment, patients are followed at 3, 6, and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer

  * Locally advanced (stage III) disease
  * Unresectable disease
* Candidate for concurrent definitive chemotherapy and thoracic radiotherapy, as determined by the treating physician
* No malignant pleural effusion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* AST or ALT ≤ 2 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* FEV_1 > 600 cc
* Not pregnant or nursing
* Negative pregnancy test
* No weight loss > 10% within the past 6 months
* No known HIV disease

PRIOR CONCURRENT THERAPY:

* No prior thoracic radiotherapy
* No prior HIV protease inhibitors
* More than 5 years since prior chemotherapy
* At least 3 weeks since prior exploratory thoracotomy
* No concurrent medications that would preclude nelfinavir administration, including any of the following:

  * Amiodarone
  * Quinidine
  * Rifampin
  * Dihydroergotamine
  * Ergonovine
  * Ergotamine
  * Methylergonovine
  * Hypericum perforatum (St. John's wort)
  * Lovastatin
  * Simvastatin
  * Pimozide
  * Midazolam
  * Triazolam

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Maity, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rengan R, Mick R, Pryma DA, Lin LL, Christodouleas J, Plastaras JP, Simone CB 2nd, Gupta AK, Evans TL, Stevenson JP, Langer CJ, Kucharczuk J, Friedberg J, Lam S, Patsch D, Hahn SM, Maity A. Clinical Outcomes of the HIV Protease Inhibitor Nelfinavir With Concurrent Chemoradiotherapy for Unresectable Stage IIIA/IIIB Non-Small Cell Lung Cancer: A Phase 1/2 Trial. JAMA Oncol. 2019 Oct 1;5(10):1464-1472. doi: 10.1001/jamaoncol.2019.2095. PMID 31436839
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Nelfinavir
  cisplatin
  etoposide
  nelfinavir mesylate
  protein expression analysis
  immunohistochemistry staining method
  laboratory biomarker analysis
  biopsy
  radiation therapy
Period: Overall Study
Arm/Group | Single Arm
Started | 55
Completed | 52
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity
Description: Any grade III or higher toxicity during chemoradiation, per CTCAE
Time Frame: 90 days
Measure: Number; unit: Dose-limiting toxicities
Arm/Group | Single Arm
Number analyzed (Participants) | 55
Dose-limiting toxicities | 0

2. Primary Outcome: Maximum Tolerated Dose of Nelfinavir
Description: As determined by dose escalation rules
Time Frame: 90 days
Measure: Number; unit: mg PO twice daily
Arm/Group | Single Arm
Number analyzed (Participants) | 55
mg PO twice daily | 1250

3. Secondary Outcome: Clinical Response of Tumor
Description: Tumor size as determined by imaging
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 55
percentage of participants | 94 [86 to 100]

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/55
Serious Adverse Events (participants affected / at risk) | 21/55
Other Adverse Events (participants affected / at risk) | 40/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=55)
ANC (Blood and lymphatic system disorders) | 3 (4)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Decreased ANC (Blood and lymphatic system disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diffuse Muscle Pain (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection, Anal/perianal (Infections and infestations) | 1 (1)
Infection, Lung (pneumonia) (Infections and infestations) | 2 (2)
Leukocytes (Blood and lymphatic system disorders) | 9 (12)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenic Fever (General disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 2 (4)
Pain in extremity (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=55)
ANC (Blood and lymphatic system disorders) | 4 (12)
AST Transaminase (Blood and lymphatic system disorders) | 1 (1)
Abdominal Pain (General disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (2)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 4 (4)
Alkalosis (Metabolism and nutrition disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Altered Taste (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 24 (41)
Anxiety (Psychiatric disorders) | 8 (10)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 1 (1)
Blurred Vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis at hangnail (Infections and infestations) | 1 (1)
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Chills (General disorders) | 2 (2)
Cholesterol (Metabolism and nutrition disorders) | 1 (1)
Confusion / Forgetfulness (Nervous system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 26 (42)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (28)
Cramping (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 3 (7)
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased ALC (Blood and lymphatic system disorders) | 1 (5)
Decreased ANC (Blood and lymphatic system disorders) | 10 (17)
Decreased Albumin (General disorders) | 1 (1)
Decreased Leukocytes (Blood and lymphatic system disorders) | 4 (11)
Decreased Magnesium (General disorders) | 2 (4)
Decreased Platelets (Blood and lymphatic system disorders) | 4 (4)
Decreased WBC (Blood and lymphatic system disorders) | 4 (5)
Decreased hemoglobin (Blood and lymphatic system disorders) | 5 (11)
Decreased leukocytes (Blood and lymphatic system disorders) | 6 (13)
Decreased platelets (Blood and lymphatic system disorders) | 3 (5)
Dehydration (Gastrointestinal disorders) | 22 (34)
Depression (Psychiatric disorders) | 9 (11)
Dermatitis (Skin and subcutaneous tissue disorders) | 6 (7)
Dermatitis radiation (Injury, poisoning and procedural complications) | 8 (12)
Desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 24 (45)
Difficulty Swallowing (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 12 (14)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 16 (29)
Dysphagia (Gastrointestinal disorders) | 22 (38)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (23)
Dysuria (Renal and urinary disorders) | 1 (1)
Esophagitis (Infections and infestations) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 6 (6)
Epigastrum (General disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Esophageal Pain (General disorders) | 8 (10)
Esophagitis (Gastrointestinal disorders) | 34 (63)
Facial Erythema (General disorders) | 1 (1)
Fatigue (General disorders) | 33 (71)
Feet Tingling (General disorders) | 1 (1)
Fever (General disorders) | 6 (8)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flushing (Blood and lymphatic system disorders) | 1 (1)
Other GI (Gastrointestinal disorders) | 3 (3)
Giddiness (General disorders) | 1 (1)
Hand Laceration (Injury, poisoning and procedural complications) | 1 (1)
Hand Tremors (General disorders) | 1 (1)
Headache (General disorders) | 9 (10)
Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Heart palpitations / A-fib / Chest pains (Cardiac disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 8 (9)
Heavy chest (General disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 25 (70)
Hemoptysis (Blood and lymphatic system disorders) | 4 (5)
Hemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Hiccups (General disorders) | 2 (3)
Hoarseness (General disorders) | 7 (7)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 4 (4)
Hypercalcemia (Blood and lymphatic system disorders) | 2 (2)
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 26 (80)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (7)
Hyperpigmentation in RT Field (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 (66)
Hypoantremia (General disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 26 (57)
Hypoglycemia (Blood and lymphatic system disorders) | 8 (12)
Hypokalemia (Blood and lymphatic system disorders) | 16 (26)
Hypomagnesemia (Blood and lymphatic system disorders) | 9 (20)
Hyponatremia (Blood and lymphatic system disorders) | 31 (62)
Hypotension (Cardiac disorders) | 8 (9)
Increased ALT (Endocrine disorders) | 6 (6)
Increased Alk Phosphates (Blood and lymphatic system disorders) | 4 (5)
Increased Creatinine (Blood and lymphatic system disorders) | 2 (2)
Increased DOE (General disorders) | 1 (1)
Increased Triglycerides (Blood and lymphatic system disorders) | 1 (1)
Infected L Eye (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9)
Intermittent Decreased Magnesium (Blood and lymphatic system disorders) | 1 (1)
Irregular Menses (Reproductive system and breast disorders) | 1 (1)
Jaw Pain (General disorders) | 1 (1)
Joint pain (General disorders) | 1 (2)
L Arm Pain (General disorders) | 1 (1)
LLE DVT (Blood and lymphatic system disorders) | 1 (1)
Left bundle branch block (Cardiac disorders) | 1 (1)
Left side burning sensation (General disorders) | 1 (1)
Leg Cramps (General disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 24 (72)
Leukopenia (Blood and lymphatic system disorders) | 1 (3)
Light headedness (General disorders) | 1 (1)
Loose Stool (Gastrointestinal disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 5 (16)
decreased total protein (Metabolism and nutrition disorders) | 2 (2)
Mood Alteration (Psychiatric disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 30 (59)
Neck Swelling (General disorders) | 1 (1)
Neuropathy (General disorders) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 9 (19)
Night Sweats (General disorders) | 2 (2)
Nosebleed (General disorders) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 4 (5)
Oral Mucositis (Infections and infestations) | 1 (1)
Orthostatic Hypotension (Blood and lymphatic system disorders) | 8 (8)
Pain (General disorders) | 8 (8)
Palmar Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pancytopemia (Blood and lymphatic system disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Pharyngeal hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 12 (29)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Poor bladder function (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
R Thoracic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rad Derm (Skin and subcutaneous tissue disorders) | 2 (3)
Radiation Dermatitis (Injury, poisoning and procedural complications) | 5 (9)
Radiation recall reaction (dermatologic) (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Rectal Pain 2d Herpes (Reproductive system and breast disorders) | 1 (1)
Reflux (Gastrointestinal disorders) | 3 (3)
Respiratory Infection (Infections and infestations) | 1 (1)
SOB (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Salivary Gland Changes (Gastrointestinal disorders) | 1 (1)
Severe headache (General disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Rash / Dryness (XRT Derm) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Sensation - burning (Skin and subcutaneous tissue disorders) | 1 (1)
Skin in rad portal (Skin and subcutaneous tissue disorders) | 1 (1)
Sleepiness (General disorders) | 1 (1)
Sore R Cheek in Mouth (General disorders) | 1 (1)
Sore Throat (Gastrointestinal disorders) | 4 (4)
Stomach cramping (Gastrointestinal disorders) | 2 (2)
Stye (Eye disorders) | 1 (1)
Suprapubic Pain 2d UTI (Renal and urinary disorders) | 1 (1)
Sweating (General disorders) | 3 (3)
Swelling of Ankles (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Systolic Blood Pressure (Cardiac disorders) | 1 (1)
Tachycardia - A-fib (Cardiac disorders) | 1 (1)
Taste Alteration (Gastrointestinal disorders) | 3 (3)
Throat pain (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (10)
Thrush (Gastrointestinal disorders) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 8 (9)
Tunnel Vision (Eye disorders) | 1 (1)
Upper Abdominal Pain (General disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Voice Change (General disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 12 (17)
WBC Decreased (Blood and lymphatic system disorders) | 1 (4)
Weakness (General disorders) | 2 (2)
Weight Gain (General disorders) | 2 (2)
Weight Loss (General disorders) | 23 (34)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
XRT Dermatitis (Skin and subcutaneous tissue disorders) | 8 (9)
Full extravasation - AC fossa (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes